CLINICAL TRIAL: NCT01889771
Title: A Cost-effectiveness Study of Nicotine Patches Distributed Through a Quitline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-0757
Record Dates: First submitted 2013-06-14; First posted 2013-06-28 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Patch (4 weeks) (Experimental): participants receive one 4-weeks supply of nicotine patches
  Interventions: Drug: Nicotine Patch
- Nicotine Patch (8 weeks) (Experimental): participants receive up to 8 weeks of nicotine patches in up to two 4-week supplies
  Interventions: Drug: Nicotine Patch

INTERVENTIONS:
Drug: Nicotine Patch — nicoderm patches are distributed in two different supplies through a telephone quitline
  Other Names: Nicoderm Committed Quit patches

SUMMARY:
The study is to understand whether distribution of two different supplies of nicotine patches through a telephone quitline has an effect on quit rates. The two different supplies are four vs. eight (in two separate four-week mailings) weeks of nicotine patches. The hypothesis is that eight weeks will be slightly more efficacious but four weeks will be more cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* All callers to the Colorado QuitLine who report currently smoking 16-20 cigarettes
* who enroll in QuitLine services
* who do not require physician approval to obtain nicotine replacement therapy
* who are willing to receive the nicotine patch

Exclusion Criteria:

* Contraindications to receiving the nicotine patch through the QuitLine without physician approval include: history of hearth disease (heart attack, chest pain, or coronary artery disease), high blood pressure, pregnancy, skin conditions such as difficult to manage psoriasis or eczema, or history of a local reaction to the nicotine patch
* those who do not complete the call in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1495 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
7-day smoking abstinence | 7 days
6-month smoking abstinence | 6 months
cost-effectiveness | 6 months
  cost per quit of each study arm will be calculated based on the total costs of the intervention from actual utilization data (nicotine patch costs + counseling call costs) and quit rates

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Burns, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Burns EK, Hood NE, Goforth E, Levinson AH. Randomised trial of two nicotine patch protocols distributed through a state quitline. Tob Control. 2016 Mar;25(2):218-23. doi: 10.1136/tobaccocontrol-2014-051843. Epub 2014 Nov 21. PMID 25416755